CLINICAL TRIAL: NCT06616207
Title: Efficacy and Safety of Topical 10% Povidone-Iodine in Preventing White Spots During Orthodontic Treatment
Brief Title: Topical 10% Povidone-Iodine in Preventing White Spots
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Greg Huang, Professor: Orthodontics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00019955; STUDY00019955 (Other: University of Washington, Human Subjects Division); Protocol #20241690 (Other: WCG IRB)
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-08

CONDITIONS: White Spot Lesions; Gingival Inflammation and Bleeding
Keywords: Povidone-Iodine; White spot lesion; Topical application of 10% Povidone- Iodine in preventing white spots; Topical 10% Povidone-Iodine In Preventing White Spots During Orthodontic Treatment
MeSH Terms: conditions — Gingivitis; Hemorrhage

STUDY DESIGN:
Intervention Model Description: In triple blind parallel interventional study model, two or more groups of participants are treated simultaneously but separately, with an intervention group (10% povidone-iodine) and placebo (double distilled water colored to match the Povidone-Iodine solution in color and taste)and will be randomly assigned at the recruitment. The researchers compare the results between the groups to see if the intervention has a preventive effect. All three parties, participants, researcher, and data analyst are unaware of who is receiving which treatment between intervention and placebo to produce the most unbiased and reliable results.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The manufacturer of Povi-One will provide the placebo. The products will be identical in appearance. Povi-One and placebo will be supplied every 6 months and stored at room temperature in locked storage in the orthodontics clinic. Povi-One and placebo will be delivered to the clinic site by the manufacturer marked with the different treatment codes. The study biostatistician will assign the codes and keep the key. The manufacturer will retain treatment codes until after analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (double distilled water matched in color and taste) will be applied
  Interventions: Drug: Placebo
- Povidone-iodine solution (Experimental): 10% Povidone and Iodine will be applied
  Interventions: Drug: Povidone-iodine solution

INTERVENTIONS:
Drug: Placebo — Placebo (Double distilled water matched in color and taste) will be applied topically by the graduate student to all tooth surfaces at the consultation appointment before the placement of fixed appliances and at 3, 6, and 9 months after appliance placement.
  Arms: Placebo
Drug: Povidone-iodine solution — Povidone-iodine solution will be applied topically by the graduate student to all tooth surfaces at the consultation appointment before the placement of fixed appliances and at 3, 6, and 9 months after appliance placement.
  Arms: Povidone-iodine solution

SUMMARY:
The goal of this clinical trial is to learn if topical application on the all surface of 10% Povidone Iodine (Povi-One) in healthy participants in transitional or permanent dentition (10-17 y) prevents new white spot lesions in the maxillary anterior teeth at 1 year of follow-up.

Researchers will compare Povi-One to a placebo to see if Povi-One works to prevent new white spot lesions.

It will also learn about the safety of topical 10% Povidone Iodine.

The main questions it aims to answer are:

1. Does Povi-One prevent the development of any white spot lesion on the surface of maxillary anterior teeth?
2. Does Povi-One lower the probability of any International Caries Detection and Assessment System (ICDAS) score greater than 0 and mean modified Löe-Silness Gingival Index (GI) in the intervention group?

Researchers will

1. Score GI without cleaning participants teeth, then score ICDAS of maxillary and mandibular incisors after participants brush and floss their teeth and take a photograph of maxillary 6 anterior teeth
2. Apply Povi-one (or control) at the consultation appointment before placing fixed orthodontic appliances and 3, 6, and 9 months after appliance placement

Researchers will

1. Recall using Zoom 24-48 hours after the first application of Povi-One and examine the participant's mouth for oral lesions using a structured paper checklist
2. Interview the caregiver to complete a paper questionnaire on adverse effects

Researchers will

1. Score GI, and then score ICDAS of maxillary and mandibular incisors in 6, 12 months after appliance placement
2. Evaluate the development of white spot lesions on maxillary central and lateral incisors in 6, and 12 months after appliance placement

DETAILED DESCRIPTION:
Protocol:

Efficacy and Safety Of Topical 10% Povidone-Iodine In Preventing White Spots During Orthodontic Treatment

Design:

A triple-blind randomized trial with two arms (10% Povidone Iodine, Placebo) where the primary outcome is the percentage of patients with at least one new white spot lesion on the maxillary anterior teeth at 1 year of follow-up. The secondary outcomes will utilize the ICDAS on the upper and lower anterior teeth, a modified Gingival Index, and Acceptability.

Hypothesis:

Participants treated with the test agent will be less likely to develop any enamel decalcification than participants treated with the placebo comparator. Also, the probability of any ICDAS score greater than 0 and mean modified Gingival Index will be lower in the treatment group than in the comparator.

Recruitment/Consent:

The participants will be recruited as they begin treatment. The orthodontic graduate student will briefly present the study and ask if the child/teen and caregiver (parent, guardian) are willing to talk about the study and then, if the child/teen and caregiver are willing, a research assistant will further explain participation and gain informed assent from the child/teen and consent from the parent.

Intervention:

Povi-One (10% povidone-iodine) will be applied topically by the graduate student to all tooth surfaces at the consultation appointment (baseline) before the placement of fixed appliances. Povi-one (or control) will be applied again at 3, 6, and 9 months after appliance placement by the graduate student.

Control:

The placebo (double distilled water colored to match the Povidone-Iodine solution in color and taste) application procedure is identical to that of the test product. The manufacturer will provide the placebo.

Concomitant Treatment:

No change will be made in orthodontic treatment. Any application of fluorides or other dental treatment will be recorded from the EHR. The participant and/or caregiver will be asked whether the participant is using any OTC fluoride products or had any fluoride applied by their dentist.

Management of agents (Povi-One and placebo) Povi-One and placebo will be delivered to the clinic site by the manufacturer marked with the different treatment codes. Treatment codes will be retained by the manufacturer until after analysis. Fresh products will be supplied every 6 months and stored at room temperature in locked storage in the orthodontics clinic.

Retention:

The drop-out rate of patients in the graduate orthodontic clinic once treatment begins is less than 5%

Sample size determination:

The sample size is based on recent data collected on adolescent patients in the UW graduate orthodontic clinic. Assuming a 50% incidence of any new white spot lesions, as identified by intra-oral photographs at 12 months in the placebo sample, and a reduction of 60% in the test sample, the sample size based on a two-sample chi-square test using a 0.05 significance level and 80% power is 39 participants per group (78 total) without accounting for attrition. Assuming 5% attrition at 12 months, the sample size required is 41 per group (82 total). Assuming an 80% acceptance rate and about 125 new patients in the required age range per year at the UW graduate orthodontic clinic, the sample of 80 patients can be accrued in one 1 year.

Data Management:

The demographic data, clinical evaluation data, and post-treatment reports will be recorded on paper forms precoded with the participant ID. These forms will be collected and kept in a locked file until entered into a computer database. The photographic images will be identified by participant ID and date and uploaded to a secure study computer.

Analysis:

The analysis will be based on the intention-to-treat principle. Binary outcomes will be summarized for each study arm and time point by frequency and percentage and quantitative outcomes will be summarized by mean, standard deviation, median, interquartile range, and range. A chi-square test will be used to compare the percentage of patients in each group that develop at least one new white spot lesion. A chi-square will be also used to compare the incidence of any ICDAS score greater than 0 and a two-sample test will be used to compare the mean modified Gingival Index and Acceptability. If the distribution of the modified Gingival Index or Acceptability is skewed, a non-parametric Mann-Whitney U test will be used. Log-linear regression with robust standard errors will used to compare the number of new ICDAS scores greater than 0 if sufficient numbers of participants have more than 1 new lesion (Hardin et al., 2003). If the attrition is greater than 10% at 12 months, multiple imputation methods will be used to account for the missing data and maintain the intention-to-treat analysis (Rubin et al., 1987). All analysis will be performed using R Version 4.3.0 (R Core Team, 2023).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and teens (10-17 years old)
* Transitional or permanent dentition of at least 4 permanent anterior teeth in each arch
* Full fixed appliance orthodontic treatment is expected to last at least one year

Exclusion Criteria:

* Allergies to iodine
* Chronic prophylactic use of antibiotics
* Diagnosis of thyroid disease
* Conditions that could impair routine oral hygiene procedures.
* Pregnant at enrollment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Photograph | From enrollment (baseline) to the 12 months after the placement of fixed appliances
  6 maxillary anterior teeth (central incisors, lateral incisors, and canines) will be photographed with a clinical cam in a 10-degree tilted head position to reduce reflection without drying teeth. A new development of white spot lesion of the maxillary 4 anterior teeth using a photograph at a baseline (before the placement of fixed appliances). The images will be labeled with randomly assigned patient ID numbers and dates, and stored on a password-protected computer for later analysis. The orthodontic graduate students will be trained to label the photos, and then deliver them to the study coordinator. A trained and calibrated independent evaluator will assess whether there are new white spot lesions by comparing progress with the baseline photos taken before the placement of fixed appliances. The examiner will be blind to group assignments.

SECONDARY OUTCOMES:
Gingival index | From enrollment (baseline) to the 12 months after the placement of fixed appliances
  The gingival index will be evaluated at the baseline (before the placement of the fixed appliances, 6 months, and 12 months after the placement) Scoring gingival index will be performed before the patient performs any oral hygiene procedures at the time of the visit. A modification of the Löe-Silness Gingival Index (GI) will be used, scoring the mid-labial aspect of the gingiva of each anterior tooth on a scale from 0 (normal gingiva); 1 (Mild inflammation: slight change in color and slight edema but no bleeding on probing); 2 (Moderate inflammation: redness, edema, and glazing, bleeding on probing); to 3 (severe inflammation: marked redness and edema, ulceration with tendency to spontaneous bleeding). Orthodontic graduate students will receive training and complete a calibration exercise for scoring the GI.
International Caries Detection and Assessment System (ICDAS) | From enrollment (baseline) to the 12 months after the placement of fixed appliances
  After the gingival index has been completed, patients will be asked to brush and floss their teeth, and any residual plaque can be removed with a micro brush.
  ICDAS will be evaluated at the baseline (before the placement of the fixed appliances, 6 months, and 12 months after the placement). Regarding the ICDAS, only the anterior teeth will be assessed clinically by the graduate orthodontic student. No magnification will be used. The graduate student examiners will be trained and calibrated to establish inter-rater reliability on a sample of 10 patients with and without ICDAS pre-cavitated lesions by a trained gold standard examiner . (Minimum acceptable ICC=.7) A review for examiners will be held for 1 year.

OTHER OUTCOMES:
Visual analog scale (VAS) | From enrollment (baseline) to the 12 months after the placement of fixed appliances
  After the first topical application in the clinic, the participant will complete a 100 mm VAS anchored with "not acceptable at all" to "completely acceptable." This assessment will be completed again at the three-month recall.
Safety measure (allergic reaction and adverse effect) | From enrollment (baseline) to the 12 months after the placement of fixed appliances
  Participants will be recalled by the orthodontic graduate students using Zoom 24-48 hours after the first application and the participant's mouth will be examined for oral lesions using a structured paper checklist which will include the participant ID, date, and the name of the person completing the checklist.
  At the same appointment, the caregiver will be interviewed to complete a paper questionnaire on adverse effects. The orthodontic graduate students will interview the caregiver who is self-identified as the main adult responsible for the participants' orthodontic care.
  Caregiver and participants will be given an emergency telephone number and asked to report significant abnormalities the participant experiences. The principal investigator will review and follow up. If the patient is having a severe medical emergency, they will be directed to contact their physician and/or go to the emergency room immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Huang, DMD, MSD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, School of Dentistry Department of Orthodontics, 1959 NE Pacific St. Health Sciences Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Sharing IPD will be restricted or carefully managed to ensure participants safety. Researchers have ethical obligations to protect the participants. When individuals agree to participate in a trial, they often do so with the understanding that their personal data will remain confidential. Also, Participants may not have given explicit consent for their data to be shared beyond the scope of the specific clinical trial. Especially in this trial, participants are children and teenagers under 18 considered a vulnerable population in clinical trials, so additional precautions are taken to ensure their safety and privacy. Protecting the individual participant data of minor participants in clinical trials is crucial due to their vulnerable status, the legal requirements, and the potential for harm that could arise from breaches in privacy or confidentiality.

REFERENCES:
- [Background] Sundararaj D, Venkatachalapathy S, Tandon A, Pereira A. Critical evaluation of incidence and prevalence of white spot lesions during fixed orthodontic appliance treatment: A meta-analysis. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):433-9. doi: 10.4103/2231-0762.167719. PMID 26759794
- [Background] Julien KC, Buschang PH, Campbell PM. Prevalence of white spot lesion formation during orthodontic treatment. Angle Orthod. 2013 Jul;83(4):641-7. doi: 10.2319/071712-584.1. Epub 2013 Jan 4. PMID 23289733
- [Background] Buschang PH, Chastain D, Keylor CL, Crosby D, Julien KC. Incidence of white spot lesions among patients treated with clear aligners and traditional braces. Angle Orthod. 2019 May;89(3):359-364. doi: 10.2319/073118-553.1. Epub 2018 Dec 17. PMID 30556747
- [Background] Sharab L, Loss C, Jensen D, Kluemper GT, Alotaibi M, Nagaoka H. Prevalence of white spot lesions and gingival index during orthodontic treatment in an academic setting. Am J Orthod Dentofacial Orthop. 2023 Jun;163(6):835-842. doi: 10.1016/j.ajodo.2022.08.023. Epub 2023 Jan 29. PMID 36720655
- [Background] Richter AE, Arruda AO, Peters MC, Sohn W. Incidence of caries lesions among patients treated with comprehensive orthodontics. Am J Orthod Dentofacial Orthop. 2011 May;139(5):657-64. doi: 10.1016/j.ajodo.2009.06.037. PMID 21536209
- [Background] Lucchese A, Gherlone E. Prevalence of white-spot lesions before and during orthodontic treatment with fixed appliances. Eur J Orthod. 2013 Oct;35(5):664-8. doi: 10.1093/ejo/cjs070. Epub 2012 Oct 8. PMID 23045306